CLINICAL TRIAL: NCT01617460
Title: A Long-term Administration Study of Aripiprazole in Children and Adolescents (Age: 6 to 17 Years) With Autistic Disorder
Brief Title: A Long-term, Extended Treatment Study of Aripiprazole in Pediatric Patients With Autistic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-11-003
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Autistic Disorder
Keywords: Autistic Disorder, children and adolescents; aripiprazole; Long-term safety study; children and adolescents
MeSH Terms: conditions — Autistic Disorder | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): administered orally once daily
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Flexibly dose administered orally once daily

SUMMARY:
The objective of this study is to investigate the safety and efficacy of aripiprazole orally administered over long term in subjects who complete a short-term treatment study of pediatric Autistic Disorder (031-11-002 study).

ELIGIBILITY:
Inclusion Criteria:

* The patient meets Autistic disorder diagnostic criteria defined in DSM-IV-TR.
* The patient has completed the 031-11-002 study (the patient has visited the hospital during week8)
* Inpatient or outpatient status

Exclusion Criteria:

* The patient is currently diagnosed with another disorder on the autism spectrum in DSM-IV-TR, including Asperger's, Rett's Disorder, PDD-NOS, Childhood Disintegrative Disorder, or Fragile-X Syndrome.
* Patients who fall under a contraindication listed in the ABILIFY package insert
* Others

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2012-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - Chubu Region
  - Chugoku Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region

REFERENCES:
- [Derived] Ichikawa H, Hiratani M, Yasuhara A, Tsujii N, Oshimo T, Ono H, Tadori Y. An open-label extension long-term study of the safety and efficacy of aripiprazole for irritability in children and adolescents with autistic disorder in Japan. Psychiatry Clin Neurosci. 2018 Feb;72(2):84-94. doi: 10.1111/pcn.12607. Epub 2017 Nov 8. PMID 28941259

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Aripiprazole was orally administered once daily to the subjects who completed the 031-11-002 study until the new indication of irritability in pediatric autistic disorder was approved, if not discontinued.
  The starting dose was 1 mg/day, and the dose was escalated to 3, 6, 9, 12, and 15 mg/day in a stepwise manner.
Period: Overall Study
Arm/Group | Aripiprazole
Started | 86
Completed | 46
Not Completed | 40
Not completed — Adverse Event | 10
Not completed — Physician Decision | 16
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 69
Region of Enrollment [Number; unit: participants]
  Japan | 86

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at the Final Assessment in Aberrant Behavior Checklist Japanese Version (ABC-J) Irritability Subscale Score
Description: The ABC-J Irritability subscale consists of 15 items. Each item scores range from 0 to 3: 0 = No problem, 1 = Mild aberrant behavior, 2 = Moderate aberrant behavior, and 3 = Severe aberrant behavior. Individual scores were summed, therefore, the overall score range was between 0-45. Higher scores represent worse condition.
Time Frame: Baseline, the final administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 86
units on a scale | -3.2 (8.1)

ADVERSE EVENTS:
Time Frame: From the start date of investigational medicinal product (IMP) administration to date of the final examination
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 10/86
Other Adverse Events (participants affected / at risk) | 84/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=86)
Malaise (General disorders) | 1
Lymphadenitis bacterial (Infections and infestations) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Autism (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Glomerulonephritis acute (Renal and urinary disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Sexual abuse (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=86)
Conjunctivitis allergic (Eye disorders) | 5
Dental caries (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 6
Salivary hypersecretion (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 12
Pyrexia (General disorders) | 8
Bronchitis (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 10
Influenza (Infections and infestations) | 25
Nasopharyngitis (Infections and infestations) | 53
Pharyngitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 8
Arthropod bite (Injury, poisoning and procedural complications) | 5
Contusion (Injury, poisoning and procedural complications) | 6
Weight increased (Investigations) | 21
Increased appetite (Metabolism and nutrition disorders) | 10
Decreased appetite (Metabolism and nutrition disorders) | 7
Autism (Nervous system disorders) | 5
Headache (Nervous system disorders) | 5
Somnolence (Nervous system disorders) | 28
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9
Eczema (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No